CLINICAL TRIAL: NCT04134689
Title: DOT Selfie: A Mobile Health Intervention With Transfer of Social Bundle Incentives to Increase Treatment Adherence in Tuberculosis Patients in Uganda: A Randomized Control Trial.
Brief Title: DOT Selfie: A Mobile Technology Intervention to Evaluate Treatment Adherence Among Tuberculosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: Makerere University (Other)
Responsible Party: Principal Investigator, Juliet Nabbuye Sekandi, Assistant Professor, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PROJECT00000571
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Tuberculosis
Keywords: Tuberculosis,; Video Directly Observed Treatment; Directly Observed Treatment; Uganda; Treatment adherence; mHealth
MeSH Terms: conditions — Tuberculosis; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: This is an open-label parallel pilot RCT where adult male and female patients with a new diagnosis of TB (N=144) will be randomized to DOT selfie (n=72) and standard in-person DOT (n=72). Patients in the DOT selfie arm will receive the intervention, which will comprise a smart phone, the VDOT App, a prepaid weekly internet bundle and text message medication reminders. Patients receiving sin-person DOT will serve as the control arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DOT Selfie Intervention Arm (Active Comparator): The DOT Selfie Intervention will comprise a smart phone, the VDOT App, a prepaid weekly internet bundle and text message medication reminders.
  Patients in this arm will receive detailed training (in English or Luganda) on VDOT use prior to starting treatment. Each patient will be required to record and submit daily videos as they self-administer their medication. Patients who successfully submit their videos for seven consecutive days will receive a weekly incentive in the form of social bundles of airtime minutes. A prepaid internet bundle will also be uploaded to each mobile phone weekly to allow for daily video uploads. Additionally, patients will receive text message medication reminders to encourage treatment compliance.
  Interventions: Device: DOT Selfie Intervention
- In-person DOT Control Arm. (Active Comparator): Patients in this arm will be managed according to the usual clinical practice in Uganda i.e. community- or home-based directly observed treatment .Patients in this arm will make prior arrangements with a study nurse to determine a convenient meeting place (e.g. at the patient's work, home etc.) The study nurse will then meet the patient at this location. At each daily meeting, the patient will self-administer the TB drugs as the study nurse directly observes and documents (date, time, drug dosing etc.) At the end of each meeting, the patient and nurse will agree on a convenient meeting place for the next day's dosing. These daily meetings will continue until treatment completion. The study nurse will record patient's medication intake, as well as the time taken to reach the patient, amount of money spent on round-trip transportation, and total amount of time spent during each patient encounter.
  Interventions: Other: In-person DOT

INTERVENTIONS:
Device: DOT Selfie Intervention — This comprises a smart phone, the VDOT App, a prepaid weekly internet bundle and text message medication reminders
  Other Names: VDOT (Video Observed Treatment)
  Arms: DOT Selfie Intervention Arm
Other: In-person DOT — Directly observed TB treatment by a health-worker either in a patient's home or at an agreed upon location within the community.
  Other Names: Standard DOT
  Arms: In-person DOT Control Arm.

SUMMARY:
This is a randomized controlled trial (RCT) to determine whether Video Observed Treatment (VDOT) using social internet bundle incentives for tuberculosis (TB) is an effective way to improve medication adherence in TB treatment, compared with standard in-person treatment (home-/ community-based).

The study will include two study arms: one will receive TB treatment using the standard in-person DOT, and the other through VDOT. All patients (regardless of study arm) will receive daily TB treatment under home- or community-based observation . For patients in the In-person DOT arm, this will be observed and recorded daily by a study nurse. Patients in the VDOT arm however, will be required to record and upload their daily medication intake using a mobile phone App. As a form of incentive, these patients will be rewarded with social internet bundles for every 7 consecutive video uploads. Additionally, they will be sent motivational text messages to encourage treatment compliance.

Regardless of study arm, all patients will have 2,4, and 6 monthly clinic visits for clinical and/or sputum assessments. Each patient will also complete a Morisky Medication Adherence Scale (MMAS) questionnaire at treatment completion.

DETAILED DESCRIPTION:
Eligible patients will be randomised in equal proportions between the DOT Selfie Intervention and In-person DOT Control arms. All patients will self-administer TB drugs daily for 6 months, or as prescribed by their physician. Once recruited, all patients will receive routine education on TB treatment, side-effects and the importance of adherence. They will also receive a baseline survey to collect data on demographics, personal, social and clinical characteristics, cell phone/smartphone ownership and prior experience with use of video camera features. Patients will be informed that regardless of the intervention allocation, they will be required to return to the clinic for study follow up at 2, 4 and 6 months to complete a follow-up interview with study staff (clinical and/ or sputum assessments).

DOT Selfie Intervention Arm. The DOT Selfie Intervention will comprise a smart phone, the VDOT App, a prepaid weekly internet bundle and text message medication reminders. The smart phone will be equipped with a camera that supports video recording. Additionally, it will have internet access, and an operating system capable of running downloaded applications. The VDOT App is a free, downloadable, passcode-protected mobile App provided by SureAdhere. It is equipped with video recording features and automatic, encrypted, time-stamped video uploads to a secure server. This enables patients to securely and confidentially document each medication dose taken. The VDOT system has a feature to adapt and personalize text messages either in English or Luganda. These text messages will include reminders for patients to take their medications, lists of common medication side effects and motivational messages to encourage patients to continue taking their medications and report any side effects.

Upon assignment to VDOT intervention arm, patients will receive detailed training (in English or Luganda) on VDOT use, using a detailed training manual provided by SureAdhere. Patients will also be trained on how to lay out each drug on a labelled laminated medication sheet with a space for each drug and take each drug type individually saying either the name of the drug or the color of the pills, size, and the number taken. Participants will be asked to show their mouth is empty by opening their mouth and sticking out their tongue and finally be asked to report any symptoms from a list of key side effects (which will be printed on the reverse of the laminated medication sheet - Appendix j). Any reported or observed side effects will be addressed by study nurses as indicated in Appendix k. Training will include watching of some test videos.

Once training is complete, the study will then begin with patients receiving the intervention (smart phone, the VDOT App, prepaid weekly internet bundle and text message medications reminders). Each patient will be required to record and submit daily videos as they self-administer their medication, when and where it works best for them. For each patient, Day 1 of the study will the mark the day the first dose of TB drugs was self-administered. Patients who successfully submit their videos for seven consecutive days will receive a weekly incentive in the form of social bundles of airtime minutes. Patients will be encouraged to try and maintain full compliance with daily drug regimen through personalized text message reminders such as "Taking your pills will help you get better and keep you from infecting family and friends." They will also be encouraged to report side effects and other related concerns through the VDOT system.

VDOT videos recorded by patients using the SureAdhere App, will be uploaded to 99DOT, a secure server and HIPAA compliant web portal used to review and track patients medication intake videos. These videos will be submitted automatically as soon as the phone is connected to a cellular data network (data plan provided with phone) or wireless network. At the clinic, a trained study nurse will log into the 99DOTs secured system via a tablet or laptop to download, review the patients' daily videos and document adherence according to a pre-specified protocol for VDOT. The nurse will view the date and time stamped videos on 99DOT, to document each medication dose taken. The nurse will thus be able to track missed videos, reported side-effects and follow-up with appropriate support advice to patients using actions specified in the study protocol. The nurse will log the time taken to contact the patient by phone, text, or in person to manage adherence problems or address any issues. VDOT videos will be read by a study nurse/VDOT observer daily during weekdays with weekend videos read on Mondays.

No incentives or travel costs will be provided but patients will be able to make use of study smartphone for e-mails, domestic telephone calls and internet searches (limited data downloads apply). Patients will be expected to return the smartphone to the clinic upon completion of their treatment.

In-person DOT Control Arm:

Patients in this arm will be managed according to usual clinical practice in Uganda. This will require prior arrangements to be made between the study nurse(s) and each patient, for a convenient meeting place (e.g. at the patient's work, home etc.) to be agreed upon. The study nurse will then be required to meet the patient daily at this location. At each daily meeting, the study nurse will provide the prescribed medication and the patient will swallow each TB medication as the study nurse directly observes and documents (date, time, drug dosing etc.) For each patient, Day 1 of the study will the mark the day the first dose of TB drugs was self-administered. Patients will be encouraged by the study nurse to report any side effects experienced, or any other related concerns. The study nurse will also encourage patients to maintain full compliance, by continuing to meet daily to have the nurse directly observe their self-administration of the drug. At the end of each meeting, the patient and nurse will agree on a convenient meeting place for the next day's dosing. The study nurse will record all of these and follow-up with appropriate support advice to manage adherence problems or other issues, using actions specified in the study protocol. The nurse will also log the time taken to reach the patient, amount of money spent on round-trip transportation, and total amount of time spent during each patient encounter.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for the trial must comply with all of the following at randomization:

1. New patients with clinically and/or microbiologically-confirmed TB or those who initiated treatment within one month (the investigators chose to enrol new cases because of lower likelihood of drug-resistant disease),
2. Age 18 to 65 years,
3. Residents of Kampala within 30 km of study clinic (to facilitate close follow-up),
4. Signed informed consent
5. Ability to speak and read Luganda or English language.

Exclusion Criteria:

1. Previous history of TB, multidrug resistant (MDR) or extensively drug-resistant (XDR) TB 2. Very ill patients 3. A cognitive or physical disability that prevents full participation in VDOT (e.g., vision, hearing, physically challenged, inability to swallow medications).

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Adherence level | 6 months
  Calculated as the number of observed doses (by videos or by a DOT worker) divided by the number of prescribed doses over the 6-month treatment period.

SECONDARY OUTCOMES:
Sputum conversion | 2, 4 and 6 months
  Proportion of patients with sputum conversion to treatment at 2, 4, and 6 months or end of treatment
Treatment completion | 6 months
  Proportion of patients completing their treatment
Clinical response | 2, 4 and 6 months
  Proportion of patients improving clinically (cough, weight gain, night sweats, fever, appetite) at 2, 4, and 6 months or end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Juliet N Sekandi, MD, MS, DrPH, Principal Investigator — University of Georgia
Locations (1):
- University of Makerere School of Public Health, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will be uploaded to the NIH portal of funded projects, in compliance with NIH requirements.

REFERENCES:
- [Background] Moore RD, Chaulk CP, Griffiths R, Cavalcante S, Chaisson RE. Cost-effectiveness of directly observed versus self-administered therapy for tuberculosis. Am J Respir Crit Care Med. 1996 Oct;154(4 Pt 1):1013-9. doi: 10.1164/ajrccm.154.4.8887600.
- [Background] Toczek A, Cox H, du Cros P, Cooke G, Ford N. Strategies for reducing treatment default in drug-resistant tuberculosis: systematic review and meta-analysis. Int J Tuberc Lung Dis. 2013 Mar;17(3):299-307. doi: 10.5588/ijtld.12.0537. Epub 2012 Dec 4. PMID 23211716
- [Background] Karumbi J, Garner P. Directly observed therapy for treating tuberculosis. Cochrane Database Syst Rev. 2015 May 29;2015(5):CD003343. doi: 10.1002/14651858.CD003343.pub4. PMID 26022367
- [Background] Mirsaeidi M, Farshidpour M, Banks-Tripp D, Hashmi S, Kujoth C, Schraufnagel D. Video directly observed therapy for treatment of tuberculosis is patient-oriented and cost-effective. Eur Respir J. 2015 Sep;46(3):871-4. doi: 10.1183/09031936.00011015. Epub 2015 Mar 18. No abstract available. PMID 25792632
- [Background] Story A, Garfein RS, Hayward A, Rusovich V, Dadu A, Soltan V, Oprunenco A, Collins K, Sarin R, Quraishi S, Sharma M, Migliori GB, Varadarajan M, Falzon D. Monitoring Therapy Compliance of Tuberculosis Patients by using Video-Enabled Electronic Devices. Emerg Infect Dis. 2016 Mar;22(3):538-40. doi: 10.3201/eid2203.151620. PMID 26891363
- [Background] Teyhen DS, Aldag M, Centola D, Edinborough E, Ghannadian JD, Haught A, Jackson T, Kinn J, Kunkler KJ, Levine B, Martindale VE, Neal D, Snyder LB, Styn MA, Thorndike F, Trabosh V, Parramore DJ. Incentives to create and sustain healthy behaviors: technology solutions and research needs. Mil Med. 2014 Dec;179(12):1419-31. doi: 10.7205/MILMED-D-14-00111. PMID 25469962
- [Background] Gibson DG, Ochieng B, Kagucia EW, Were J, Hayford K, Moulton LH, Levine OS, Odhiambo F, O'Brien KL, Feikin DR. Mobile phone-delivered reminders and incentives to improve childhood immunisation coverage and timeliness in Kenya (M-SIMU): a cluster randomised controlled trial. Lancet Glob Health. 2017 Apr;5(4):e428-e438. doi: 10.1016/S2214-109X(17)30072-4. PMID 28288747
- [Background] Moonan PK, Quitugua TN, Pogoda JM, Woo G, Drewyer G, Sahbazian B, Dunbar D, Jost KC Jr, Wallace C, Weis SE. Does directly observed therapy (DOT) reduce drug resistant tuberculosis? BMC Public Health. 2011 Jan 7;11:19. doi: 10.1186/1471-2458-11-19. PMID 21214913
- [Background] Munro SA, Lewin SA, Smith HJ, Engel ME, Fretheim A, Volmink J. Patient adherence to tuberculosis treatment: a systematic review of qualitative research. PLoS Med. 2007 Jul 24;4(7):e238. doi: 10.1371/journal.pmed.0040238. PMID 17676945
- [Background] Elbireer S, Guwatudde D, Mudiope P, Nabbuye-Sekandi J, Manabe YC. Tuberculosis treatment default among HIV-TB co-infected patients in urban Uganda. Trop Med Int Health. 2011 Aug;16(8):981-7. doi: 10.1111/j.1365-3156.2011.02800.x. Epub 2011 May 18. PMID 21585625
- [Background] Whalen CC, Nsubuga P, Okwera A, Johnson JL, Hom DL, Michael NL, Mugerwa RD, Ellner JJ. Impact of pulmonary tuberculosis on survival of HIV-infected adults: a prospective epidemiologic study in Uganda. AIDS. 2000 Jun 16;14(9):1219-28. doi: 10.1097/00002030-200006160-00020. PMID 10894287
- [Background] Guwatudde D, Zalwango S, Kamya MR, Debanne SM, Diaz MI, Okwera A, Mugerwa RD, King C, Whalen CC. Burden of tuberculosis in Kampala, Uganda. Bull World Health Organ. 2003;81(11):799-805. Epub 2004 Jan 20. PMID 14758406
- [Background] Volmink J, Garner P. Directly observed therapy for treating tuberculosis. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD003343. doi: 10.1002/14651858.CD003343.pub3. PMID 17943789
- [Background] Amuha MG, Kutyabami P, Kitutu FE, Odoi-Adome R, Kalyango JN. Non-adherence to anti-TB drugs among TB/HIV co-infected patients in Mbarara Hospital Uganda: prevalence and associated factors. Afr Health Sci. 2009 Aug 1;9 Suppl 1(Suppl 1):S8-15. PMID 20589161
- [Background] Kisambu J, Nuwaha F, Sekandi JN. Adherence to treatment and supervision for tuberculosis in a DOTS programme among pastoralists in Uganda. Int J Tuberc Lung Dis. 2014 Jul;18(7):799-803. doi: 10.5588/ijtld.13.0753. PMID 24902555
- [Background] Garfein RS, Collins K, Munoz F, Moser K, Cerecer-Callu P, Raab F, Rios P, Flick A, Zuniga ML, Cuevas-Mota J, Liang K, Rangel G, Burgos JL, Rodwell TC, Patrick K. Feasibility of tuberculosis treatment monitoring by video directly observed therapy: a binational pilot study. Int J Tuberc Lung Dis. 2015 Sep;19(9):1057-64. doi: 10.5588/ijtld.14.0923. PMID 26260824
- [Background] Pinto LM, Udwadia ZF. Private patient perceptions about a public programme; what do private Indian tuberculosis patients really feel about directly observed treatment? BMC Public Health. 2010 Jun 22;10:357. doi: 10.1186/1471-2458-10-357. PMID 20569448
- [Background] Bulage L, Sekandi J, Kigenyi O, Mupere E. The quality of tuberculosis services in health care centres in a rural district in Uganda: the providers' and clients' perspective. Tuberc Res Treat. 2014;2014:685982. doi: 10.1155/2014/685982. Epub 2014 Sep 7. PMID 25276424
- [Background] Mafigiri DK, McGrath JW, Whalen CC. Task shifting for tuberculosis control: a qualitative study of community-based directly observed therapy in urban Uganda. Glob Public Health. 2012;7(3):270-84. doi: 10.1080/17441692.2011.552067. Epub 2011 Jun 1. PMID 21360381
- [Background] Aluvaala J, Nyamai R, Were F, Wasunna A, Kosgei R, Karumbi J, Gathara D, English M; SIRCLE/Ministry of Health Hospital Survey Group. Assessment of neonatal care in clinical training facilities in Kenya. Arch Dis Child. 2015 Jan;100(1):42-7. doi: 10.1136/archdischild-2014-306423. Epub 2014 Aug 19. PMID 25138104
- [Background] Alipanah N, Jarlsberg L, Miller C, Linh NN, Falzon D, Jaramillo E, Nahid P. Adherence interventions and outcomes of tuberculosis treatment: A systematic review and meta-analysis of trials and observational studies. PLoS Med. 2018 Jul 3;15(7):e1002595. doi: 10.1371/journal.pmed.1002595. eCollection 2018 Jul. PMID 29969463
- [Background] Lukoye D, Adatu F, Musisi K, Kasule GW, Were W, Odeke R, Kalamya JN, Awor A, Date A, Joloba ML. Anti-tuberculosis drug resistance among new and previously treated sputum smear-positive tuberculosis patients in Uganda: results of the first national survey. PLoS One. 2013 Aug 1;8(8):e70763. doi: 10.1371/journal.pone.0070763. Print 2013. PMID 23936467
- [Background] Olano-Soler H, Thomas D, Joglar O, Rios K, Torres-Rodriguez M, Duran-Guzman G, Chorba T. Notes from the Field: Use of Asynchronous Video Directly Observed Therapy for Treatment of Tuberculosis and Latent Tuberculosis Infection in a Long-Term-Care Facility - Puerto Rico, 2016-2017. MMWR Morb Mortal Wkly Rep. 2017 Dec 22;66(50):1386-1387. doi: 10.15585/mmwr.mm6650a5. No abstract available. PMID 29267264
- [Background] Morris S, Miner M, Rodriguez T, Stancil R, Wiltz-Beckham D, Chorba T. Notes from the Field: Tuberculosis Control Activities After Hurricane Harvey - Texas, 2017. MMWR Morb Mortal Wkly Rep. 2017 Dec 15;66(49):1362-1363. doi: 10.15585/mmwr.mm6649a5. No abstract available. PMID 29240726
- [Background] Ngwatu BK, Nsengiyumva NP, Oxlade O, Mappin-Kasirer B, Nguyen NL, Jaramillo E, Falzon D, Schwartzman K; Collaborative group on the impact of digital technologies on TB. The impact of digital health technologies on tuberculosis treatment: a systematic review. Eur Respir J. 2018 Jan 11;51(1):1701596. doi: 10.1183/13993003.01596-2017. Print 2018 Jan. PMID 29326332
- [Background] DeMaio J, Schwartz L, Cooley P, Tice A. The application of telemedicine technology to a directly observed therapy program for tuberculosis: a pilot project. Clin Infect Dis. 2001 Dec 15;33(12):2082-4. doi: 10.1086/324506. Epub 2001 Nov 6. PMID 11698993
- [Background] Gassanov MA, Feldman LJ, Sebastian A, Kraguljac MJ, Rea E, Yaffe B. The use of videophone for directly observed therapy for the treatment of tuberculosis. Can J Public Health. 2013 May 14;104(3):e272. doi: 10.17269/cjph.104.3869. No abstract available. PMID 23823897
- [Background] Hoffman JA, Cunningham JR, Suleh AJ, Sundsmo A, Dekker D, Vago F, Munly K, Igonya EK, Hunt-Glassman J. Mobile direct observation treatment for tuberculosis patients: a technical feasibility pilot using mobile phones in Nairobi, Kenya. Am J Prev Med. 2010 Jul;39(1):78-80. doi: 10.1016/j.amepre.2010.02.018. Epub 2010 May 26. PMID 20537846
- [Background] Krueger K, Ruby D, Cooley P, Montoya B, Exarchos A, Djojonegoro BM, Field K. Videophone utilization as an alternative to directly observed therapy for tuberculosis. Int J Tuberc Lung Dis. 2010 Jun;14(6):779-81. PMID 20487619
- [Background] Wade VA, Karnon J, Eliott JA, Hiller JE. Home videophones improve direct observation in tuberculosis treatment: a mixed methods evaluation. PLoS One. 2012;7(11):e50155. doi: 10.1371/journal.pone.0050155. Epub 2012 Nov 30. PMID 23226243
- [Background] Demeester M. Cultural aspects of information technology implementation. Int J Med Inform. 1999 Dec;56(1-3):25-41. doi: 10.1016/s1386-5056(99)00036-2. PMID 10659932
- [Background] Resnicow K, Baranowski T, Ahluwalia JS, Braithwaite RL. Cultural sensitivity in public health: defined and demystified. Ethn Dis. 1999 Winter;9(1):10-21. PMID 10355471
- [Derived] Sekandi JN, Buregyeya E, Zalwango S, Nakkonde D, Kaggwa P, Quach THT, Asiimwe D, Atuyambe L, Dobbin K. Effectiveness of a Mobile Health Intervention (DOT Selfie) in Increasing Treatment Adherence Monitoring and Support for Patients With Tuberculosis in Uganda: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2025 Jan 16;13:e57991. doi: 10.2196/57991. PMID 39715573
- [Derived] Sekandi JN, Onuoha NA, Buregyeya E, Zalwango S, Kaggwa PE, Nakkonde D, Kakaire R, Atuyambe L, Whalen CC, Dobbin KK. Using a Mobile Health Intervention (DOT Selfie) With Transfer of Social Bundle Incentives to Increase Treatment Adherence in Tuberculosis Patients in Uganda: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Jan 5;10(1):e18029. doi: 10.2196/18029. PMID 32990629